CLINICAL TRIAL: NCT06765304
Title: Preconceptional Period and Transtheoretically Based Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Şerife İrem DÖNER, Research Assistant, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DönerKarahan24
Record Dates: First submitted 2024-12-20; First posted 2025-01-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Preconceptional Care; Education

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transtheoretically Based Education Model Intervention Group (Experimental)
  Interventions: Behavioral: Transtheoretical education intervention group
- Preconceptional Period Healthy Life Behaviours Classical Education Intervention Group (Experimental)
  Interventions: Behavioral: Preconceptional Period Healthy Life Behaviours Classical Education Intervention Group
- Placebo Group (Placebo Comparator)
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Transtheoretical education intervention group — The training sessions will be held over four weeks in eight consecutive sessions (two sessions per week). Each session will last 60 minutes. The content of each training module will be designed under the following headings: Week 1 - Planning, Week 2 - Preparation, Week 3 - Action, Week 4 - Sustainability.
  Arms: Transtheoretically Based Education Model Intervention Group
Behavioral: Preconceptional Period Healthy Life Behaviours Classical Education Intervention Group — Participants will be provided with eight educational modules designed for the preconception period. Training sessions will be conducted twice weekly for 60 minutes over a four-week period.
  Arms: Preconceptional Period Healthy Life Behaviours Classical Education Intervention Group
Behavioral: Placebo — No procedures will be performed on participants.
  Arms: Placebo Group

SUMMARY:
This study aims to evaluate the effectiveness of transtheoretical model (TTM)-based training provided to women with risky lifestyle behaviors during the preconceptional period. The preconceptional period is a critical time for women to modify health behaviors, as addressing these risks early can prevent adverse obstetric outcomes. TTM conceptualizes behavior change as a process and identifies distinct stages individuals progress through during this process. The study examines the impact of TTM-based interventions on improving unhealthy lifestyle behaviors in women before pregnancy.

DETAILED DESCRIPTION:
The preconceptional period is defined as 3 months before pregnancy or at least 1-2 years before the start of unprotected sexual intercourse. Many women enter the pregnancy period with risky living conditions and behaviours including pre-existing physical and behavioural health problems, exposure to teratogenic drugs or adverse environmental conditions, genetic disorders, substance use, unhealthy diet, obesity and domestic violence. It is not possible to correct these risky behaviours which cause many adverse obstetric outcomes in the early periods when pregnancy is not yet noticed. Therefore, many modifiable risky behaviours that may adversely affect outcomes during pregnancy and are difficult to change in the short term should be addressed in the pre-pregnancy period. It is recommended that educational interventions for changing behaviour should be model-based. In this way, it is easier to determine the main factors affecting behaviour, the relationships between these factors and the elements that need to be focused on more. One of the prominent theories that can be taken as a basis for behaviour modification training is the transtheoretical model. The transtheoretical model assumes that individuals go through some stages in the process of changing their health behaviours and maintaining these changes. According to this model, behaviour change is considered as a process rather than a result. One of the prominent theories that can be taken as a basis for behaviour change training is the transtheoretical model. The transtheoretical model assumes that individuals go through some stages in the process of changing their health behaviours and maintaining these changes. According to this model, behaviour change is considered as a process rather than an outcome. This model, developed by Prochaska and DiClemente (1982), basically divides the stage at which the individual is in the change of unhealthy behaviour into five stages temporally. According to this model, people change from people who have no intention to change in adopting new behaviours (pre-planning) to people who think-design to change (planning), to activists who adopt the behaviour but have not yet changed the behaviour regularly (preparation), and to maintainers who have changed the behaviour (action) and continue this behaviour regularly (maintenance). The aim of this study was to determine the effectiveness of transtheoretical model-based training given to women with risky life behaviours in the preconceptional period.

ELIGIBILITY:
Inclusion Criteria:

Volunteering to participate in the research

* Being between the ages of 18-49 and not going through menopause
* Not having problems in speaking and understanding Turkish
* To be able to read and write
* Being sexually active
* Thinking about becoming pregnant in the next 2 years
* Having the risk score determined from the 'Preconceptional Risky Life Behaviours in Women Diagnostic Scale' to be developed by the researchers

Exclusion Criteria:

* Psychiatric illness
* Having chronic diseases (diabetes, hypertension, hypothyroidism, etc.)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Status of Risky Behaviours | Measurements will be made before starting the study and 1 month after the end of the training intervention.As the score obtained from the scale increases, it will be determined that the woman has risky life behaviours in the preconceptional period.
  Preconceptional Risky Life Behaviours in Women will be measured using the Diagnostic Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No